CLINICAL TRIAL: NCT02717247
Title: Effect of Transcranial Random Noise Stimulation of Prefrontal Cortex on Craving Supply Subject Suffering From Obesity
Brief Title: Transcranial Random Noise Stimulation in Food Addiction Treatment
Acronym: tRNS-FA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the princcipal investigator went abroad
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-A00028-41
Record Dates: First submitted 2016-03-07; First posted 2016-03-23 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Overweight, Obesity and Other Hyperalimentation (E65-E68)
Keywords: tRNS; Food addiction,; Obesity; Craving; functional magnetic resonance imaging (fMRI)
MeSH Terms: conditions — Overweight; Obesity; Food Addiction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tRNS treatment (Experimental): The intervention consists in active tRNS stimulation with cathode above the left dorsolateral prefrontal cortex (DLPFC) which corresponds to the F3 location given by the 10-20 system. Anode is above the right dorsalateral prefrontal cortex (F4).
  100 (Hertz)Hz-650Hz, 2milliampere(mA), 30min, twice daily, 5 days
  Interventions: Device: Active tRNS
- Placebo tRNS treatment (Sham Comparator): The intervention consists in placebo or sham tRNS stimulation electrode are above F3 and F4. Voltage will be ramped at the begin and end of a stimulation for 30 seconds. Placebo stimulation will consist of just applying the ramps at the begin and end of the stimulation.
  Interventions: Device: Sham tRNS

INTERVENTIONS:
Device: Active tRNS — The intervention consists in active tRNS stimulation with cathode above the left dorsolateral prefrontal cortex (DLPFC) which corresponds to the F3 location given by the 10-20 system. Anode is above the right dorsolateral prefrontal cortex (F4).
  100Hz-650Hz, 2mA, 30min, twice daily, 5 days
  Arms: Active tRNS treatment
Device: Sham tRNS — The intervention consists in placebo or sham tRNS stimulation electrode are above F3 and F4. Voltage will be ramped at the begin and end of a stimulation for 30 seconds. Placebo stimulation will consist of just applying the ramps at the begin and end of the stimulation.
  Arms: Placebo tRNS treatment

SUMMARY:
Obesity is worldwide a public health problem. According to World Health Organization (WHO), overweight and obesity are the fifth death risk factor worldwide. At least 2.8 million adults die each year. Food addiction is one of the causes of obesity that may benefit from new therapeutic options.

DETAILED DESCRIPTION:
Transcranial random noise stimulation is a noninvasive brain stimulation technic. The modulation of the electrical activity of the right and left dorsolateral prefrontal cortex (DLPFC) by tRNS is able to act on the phenomenon of craving in other addictions. This allows us to make the assumption that tRNS stimulation could constitute a treatment for food addiction especially in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female or male between 18 and 65 years old
* Patients suffering from obesity, with a BMI ≥ 30.
* Food dependence score at the Yale Food addiction Scale ≥ 3

Exclusion Criteria:

* Presence of a an other psychiatric diagnosis of Axis I (DSM IV);
* Presence of addictive comorbidity other than food addiction
* Psychotropic treatment;
* Pregnancy or lactation;
* Contraindication to fMRI .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Effects on craving frequencies | Change from baseline after 3 months
  by questionnaires scores and declarative number of food

SECONDARY OUTCOMES:
change in body weight | Change from baseline after 3 months
change in waist circumference | Change from baseline after 3 months
change in body mass index | Change from baseline after 3 months
change in biological markers such as lipid profile, ghrelin, leptin, prolactin | Change from baseline after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: D'AMATO THIERRY, PUPH, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No